CLINICAL TRIAL: NCT05978960
Title: An EXErcise Regimen Designed to Improve Body Composition, Functional Capacity, and Strength After Treatment for Breast Cancer with Nutrition Optimization
Brief Title: EXERT-BCN: an Exercise and Nutrition Regimen to Designed to Improve Body Composition After Treatment for Breast Cancer
Acronym: EXERT-BCN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Responsible Party: Principal Investigator, Colin Champ, MD, Radiation Oncologist, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-131-SG
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer
Keywords: breast cancer; nutrition; body composition
MeSH Terms: conditions — Breast Neoplasms | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Resistance training with high quality low-carbohydrate nutrition regimen (Experimental): The regimen will consist of an intense resistance training program with linear progression and the goal of increase strength, mobility, muscle mass, and functional capacity. The nutrition program will avoid calorie counting, and instead focus on quality, while maximizing protein and limiting carbohydrates.
  Interventions: Other: Nutrition and resistance training exercise intervention

INTERVENTIONS:
Other: Nutrition and resistance training exercise intervention — 3 month 2-3 times/week, 60 min exercise regimen utilizes compound movements to focus on body composition, strength, and mobility. Classes are run by certified strength and conditioning specialists and adjusted for linear progression and safety, progressing from compound to isolated movements to maximize safety.
  The nutrition intervention focuses on dietary quality by following a "healthy low-carbohydrate" diet, focusing on nutrient dense foods high and avoiding processed foods and simple carbohydrates to keep totals under 100g/day. Participants will be advised to eat vegetables, avoid snacking, cook all meals with family and friends, avoid eating on the run, and focus on whole foods that require preparation. Calculations and quantification of calories will be avoided, while protein consumption goals are 1.3-1.8 g/kg per. Dietary strategy will be continuously discussed during exercise sessions and the PI will have twice monthly meetings with participants.

SUMMARY:
This protocol seeks to analyze patient outcomes of the standard of care, monitored group exercise regimen of high-load resistance training and functional exercises with compound movements in conjunction with a nutrition regimen focused on food quality under close supervision on women who have been treated for breast cancer.

DETAILED DESCRIPTION:
Excess adipose tissue is a risk factor for the diagnosis of breast cancer and is also associated with an increased risk of disease recurrence.1 Additionally weight gain during and after treatment for breast cancer is associated with a higher risk of recurrence, distant metastases, and death.2 More specifically, low muscle mass and increased adipose tissue is associated with poorer outcomes after the treatment of breast cancer.3 Yet, most women gain significant weight during and after breast cancer treatment, potentially compromising outcomes.

Effective methods to promote weight loss and improve metabolic and hormonal dysregulation, inflammation, and body composition in the breast cancer setting are urgently needed. In the noncancer setting, the promotion of high-quality diets that avoided processed food and simple carbohydrates in the DIETFITS study promoted weight loss4. However, this dietary strategy and others were utilized to result in weight loss, but do not necessarily consider maximizing body composition, i.e., muscle mass preservation or increase, and adipose tissue loss.

The major, and some would consider only, non-pharmacological method to increase muscle mass is via resistance training with an adequate stimulus and quantity to elicit and promote hypertrophy.5 Our group has already shown that profound muscle hypertrophy is attainable in a population of women undergoing treatment for breast cancer, particularly when the dose threshold of load and repetitions is met. At interim analysis, this program revealed a 2 lb. increase in muscle mass and a 6 lb. decrease in adipose tissue after a 3 month program utilizing linear progression.

Based on the DIEFITS protocol which has been described as a "healthy low-carbohydrate" diet, participants will be advised to eat nutrient dense food sources high in vitamins, minerals, and nutrients. Participants will be told to limit processed foods, sugar, bread, pasta, and other simple carbohydrates. Participants will be advised to eat plenty of colorful and nonstarchy vegetables. Finally, participants will be told to avoid snacking between meals, cook most/all meals, eat with family and friends, avoid eating food in the car or on the run, and focus on whole foods that require preparation. This protocol resulted in significant weight loss at one year. Additionally, the lack of calculations and quantification of calories leaves this as a more user-friendly option for participants.

The exercise regimen from EXERT-BC has yet to be combined with a dietary intervention. Thus, the following protocol will assess our resistance training regimen in conjunction with a nutrition intervention similar to the DIETFITS Protocol. This will allow adequate assessment of whether we can optimize body composition in these individuals with both exercise and dietary changes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-89 years
2. Women with a biopsy proven diagnosis of ductal carcinoma in situ or invasive carcinoma of the breast.
3. Women must have undergone treatment for breast cancer, including one or more of the following: surgery, radiation therapy, chemotherapy, immunotherapy, or hormonal therapy. Women undergoing active chemotherapy are not allowed on study. Treatment with targeted agents and immunotherapy is allowed.

Exclusion Criteria:

1. Any current treatment with chemotherapy for breast cancer
2. Inability to get and down off the ground or squat body weight
3. Inability to safely engage in group sessions
4. Severe arthritic, joint, cardiovascular, or musculoskeletal condition deemed by PI to be unsafe to engage in resistance training

Ages: 20 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-05-20 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2024-09-19 (Actual)

PRIMARY OUTCOMES:
Determine changes in fat mass in pounds from before to after the nutrition and exercise regimen via bioimpedance analysis | 3 months
  Measurement on bioimpedance analysis machine (Inbody 970)
Determine changes in fat mass in pounds from before to after the nutrition and exercise regimen via ultrasound | 3 months
  Measurement via ultrasound and calculation with Jackson-Pollack calculations

SECONDARY OUTCOMES:
Determine changes in bone mineral concentration in pounds from before to after the nutrition and exercise regimen | 3 months
  Measurement on bioimpedance analysis machine (Inbody 970)
Determine changes in General Anxiety Disorder-7 (GAD7) anxiety score from before to after the nutrition and exercise regimen | 3 months
  General Anxiety Disorder-7 total score for the seven questions ranges from 0 (no anxiety) to 21 (highest level of anxiety). This is calculated by assigning scores of 0 (minimum), 1, 2, and 3 (maximum), to the response categories of "not at all", "several days", "more than half the days", and "nearly every day", respectively. Higher scores mean a worse outcome.
Determine changes in Patient Health Questionnaire-9 (PHQ9) depression score from before to after the nutrition and exercise regimen | 3 months
  Patient Health Questionnaire-9 total score for the 9 questions ranges from 0 (no depression) to 27 (highest level of depression). This is calculated by assigning scores of 0 (minimum), 1, 2, and 3 (maximum), to the response categories of "not at all", "several days", "more than half the days", and "nearly every day", respectively. Higher scores mean a worse outcome.
Determine changes in EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) responses 1-5 and overall score from before to after the nutrition and exercise regimen | 3 months
  EuroQol-5 Dimensions-5 Levels total score for the 5 questions ranges from 5 (no problems on any dimension) to 25 (extreme problems on all dimensions). This is calculated by assigning scores of 1 (minimum), 2, 3, 4, and 5 (maximum), to the response categories of "no problems", "slight problems", "moderate problems", "severe problems", and "extreme problems"/"unable to", respectively. Higher scores mean worse outcomes.
Determine changes in strength via load measured in pounds from before to after the nutrition and exercise regimen | 3 months
  Load is calculated by multiplying sets by repetitions by weight lifted for a specific exercise
Determine changes in Y-balance score for each leg | 3 months
  Y-balance score adds up the distance each leg can move in the front and side directions, divided by the length of the hip. This correlates inversely with fall risk.
Determine changes in overall score of Functional Movement Screen (FMS) from before to after the nutrition and exercise regimen | 3 months
  Functional movement screen (FMS) total score for the 7 movement patterns assessed by an examiner ranges from 0 to 21. A score below 14 is felt to identify individuals at risk of injury. This is calculated by assigning scores of 0 (minimum), 1, 2, and 3 (maximum) to the response categories of "if any pain felt by the subject during the movement", "subject is unable to perform the movement", "subject performs the movement through compensatory movements", and "subject performs the movement correctly", respectively. A score below 14 is felt to identify individuals at risk of injury. Higher scores mean a better outcome.
Determine changes in resting metabolic rate in kilocalories/day from before to after the nutrition and exercise regimen | 3 months
  Measurement via VO2 Master indirect calorimeter
Determine changes in muscle mass in pounds from before to after the nutrition and exercise regimen | 3 months
  Measurement on bioimpedance analysis machine (Inbody 970)

CONTACTS AND LOCATIONS:
Locations (1):
- AHN CI Exercise Oncology and Resiliency, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Undecided at this point

REFERENCES:
- [Background] Gardner CD, Trepanowski JF, Del Gobbo LC, Hauser ME, Rigdon J, Ioannidis JPA, Desai M, King AC. Effect of Low-Fat vs Low-Carbohydrate Diet on 12-Month Weight Loss in Overweight Adults and the Association With Genotype Pattern or Insulin Secretion: The DIETFITS Randomized Clinical Trial. JAMA. 2018 Feb 20;319(7):667-679. doi: 10.1001/jama.2018.0245. PMID 29466592
- [Background] Champ CE, Carpenter DJ, Diaz AK, Rosenberg J, Ackerson BG, Hyde PN. Resistance Training for Patients with Cancer: A Conceptual Framework for Maximizing Strength, Power, Functional Mobility, and Body Composition to Optimize Health and Outcomes. Sports Med. 2023 Jan;53(1):75-89. doi: 10.1007/s40279-022-01759-z. Epub 2022 Sep 29. PMID 36175646